CLINICAL TRIAL: NCT03801239
Title: Reliability of Polish-Version Overactive Bladder Syndrom Scores (OABSS) Questionnaire and the Correlation of OABSS With the Results of UDI-6 and IIQ-7 Questionnaires
Brief Title: Reliability of Polish-Version Overactive Bladder Syndrom Scores (OABSS)
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Andrzej Wróbel, PhD, MD associated professor, Medical University of Lublin
Other Study IDs: 01/2019
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Overactive Bladder; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with Overactive Bladder (OAB): Patients completed the Polish version of the OABSS on two separate visits: Week 0 and Week 2 and additionally UDI-6, IIQ-7 during visit- Week 2.
  Interventions: Diagnostic Test: Urodynamic Study; Diagnostic Test: OABSS questionnaire fulfilment; Diagnostic Test: UDI-6 questionnaire fulfilment; Diagnostic Test: IIQ-7 questionnaire fulfilment
- patients with Mixed Urinary incontinence (MUI): Patients completed the Polish version of the OABSS on two separate visits: Week 0 and Week 2 and additionally UDI-6, IIQ-7 during visit- Week 2.
  Interventions: Diagnostic Test: Urodynamic Study; Diagnostic Test: OABSS questionnaire fulfilment; Diagnostic Test: UDI-6 questionnaire fulfilment; Diagnostic Test: IIQ-7 questionnaire fulfilment
- patients with Stress Urinary Incontinence (SUI): Patients completed the Polish version of the OABSS on two separate visits: Week 0 and Week 2 and additionally UDI-6, IIQ-7 during visit- Week 2.
  Interventions: Diagnostic Test: Urodynamic Study; Diagnostic Test: OABSS questionnaire fulfilment; Diagnostic Test: UDI-6 questionnaire fulfilment; Diagnostic Test: IIQ-7 questionnaire fulfilment

INTERVENTIONS:
Diagnostic Test: Urodynamic Study — during visit Week 0 patients had urodynamic study
Diagnostic Test: OABSS questionnaire fulfilment — during visit Week 0 and Week 2 patients fulfilled OABSS
Diagnostic Test: UDI-6 questionnaire fulfilment — during visit Week 2 patients fulfilled UDI-6 questionnaire
Diagnostic Test: IIQ-7 questionnaire fulfilment — during visit Week 2 patients fulfilled IIQ-7 questionnaire

SUMMARY:
The aim of this study was to develop and assess the effectiveness of a Polish version of OABSS and to correlate the OABSS with urodynamic study results and UDI-6, IIQ-7 questionnaires

DETAILED DESCRIPTION:
The translation into Polish followed standardized procedures. Women aged between 18-75 years were included into the study. All patients were recruited from women attending the Outpatient Clinic of the 2nd Gynecology Department of the Medical University in Lublin. SUI was observed in 290 cases; OAB in 283 patients and 249 had MUI (confirmed by medical history, and urodynamic investigation). All patients completed the Polish version of the OABSS on two separate visits: Week 0 and Week 2 and additionally UDI-6, IIQ-7 during visit- Week 2.

ELIGIBILITY:
Inclusion Criteria:

* confirmed Urinary Incontinence in Urodynamic study (SUI, OAB, MUI)
* female aged 18-75 years old

Exclusion Criteria:

* malignant disorders
* uncontrolled diabetes
* inability to understand informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were recruited from women attending the Outpatient Clinic of the 2nd Gynecology Department of the Medical University in Lublin. SUI was observed in 290 cases; OAB in 283 patients and 249 had MUI
Sampling Method: Non-Probability Sample
Enrollment: 822 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of OABSS questionnaire and Urodynamic study | 2 weeks
  Results of polish version of OABSS are correlated with Urodynamic study results

SECONDARY OUTCOMES:
Correlation of OABSS questionnaire with UDI-6 results | 2 weeks
  Results of polish version of OABSS are correlated with UDI-6 results
Correlation of OABSS questionnaire with IIQ-7 results | 2 weeks
  Results of polish version of OABSS are correlated with IIQ-7 results

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lublin, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No